CLINICAL TRIAL: NCT07209605
Title: Mini-anchor Versus Pull-out Suture for Surgical Management of Volar Plate Injuries
Brief Title: Mini-anchor Versus Pull-out Suture for Surgical Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ali Mohammed Ali Hammam, Orthopedics resident. Sohag University hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-9-19MS
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Volar Plate Injury
Keywords: Mini-anchor versus Pull-out Suture for Surgical Management of Volar Plate Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Pull-out Suture Technique (Active Comparator)
  Interventions: Procedure: Group A Pull-out Suture Technique
- Group B - Mini-anchor Technique (Active Comparator): Using the same volar approach, the volar plate will be reattached with two Mitek Micro QuickAnchors (1.3 x 3.7 mm), placed at the distal phalanx. Anchors will be inserted under fluoroscopic guidance to avoid dorsal cortex penetration. A hemimodified Kessler stitch pattern will be used with 3-0 polyester sutures.
  Interventions: Procedure: Group B- Mini-anchor Technique

INTERVENTIONS:
Procedure: Group A Pull-out Suture Technique — A Brunner volar incision will be made, and the volar plate avulsion fragment will be identified. A 2-0 nonabsorbable braided suture will be passed through the volar plate using Kessler pattern, and Keith needles will be used to exit the sutures dorsally . .
  Arms: Group A - Pull-out Suture Technique
Procedure: Group B- Mini-anchor Technique — Using the same volar approach, the volar plate will be reattached with two Mitek Micro QuickAnchors (1.3 x 3.7 mm), placed at the distal phalanx. Anchors will be inserted under fluoroscopic guidance to avoid dorsal cortex penetration. A hemimodified Kessler stitch pattern will be used with 3-0 polyester sutures.
  Arms: Group B - Mini-anchor Technique

SUMMARY:
Volar plate injuries of the joint are among the most common traumatic lesions in the hand. These injuries result from hyperextension trauma, leading to volar plate avulsion, often accompanied by collateral ligament injuries or fractures of the volar plate Conventional repair techniques include pull-out . Although widely used, pull-out sutures are associated with specific complications such as skin irritation. The external suture may also interfere with early mobilization, a key factor for good postoperative outcomes (3).

Suture anchors have emerged as a modern alternative, offering internal fixation without the need for pull out sutures. Their application is believed to promote faster recovery, minimize soft tissue irritation, and early mobilization

DETAILED DESCRIPTION:
Volar plate injuries of the joint are among the most common traumatic lesions in the hand. These injuries result from hyperextension trauma, leading to volar plate avulsion, often accompanied by collateral ligament injuries or fractures of the volar plate Conventional repair techniques include pull-out . Although widely used, pull-out sutures are associated with specific complications such as skin irritation. The external suture may also interfere with early mobilization, a key factor for good postoperative outcomes (3).

Suture anchors have emerged as a modern alternative, offering internal fixation without the need for pull out sutures. Their application is believed to promote faster recovery, minimize soft tissue irritation, and early mobilization Aim of the Work The aim of this study is to compare the clinical and functional outcomes of mini-anchor versus pull-out suture techniques in surgical management of volar plate injuries of the PIP joint.

-Place of the study: Sohag University Hospitals after approval from the institutional ethical committee.

-Type of the study: A prospective randomized clinical trial.

* Study period:

From 1/10/2025 to 1/4/2026……………

- Patients:

This study will be conducted on patients with volar plate injuries of the PIP joint. An online randomization program (http://www.randomizer.org) will be used to generate a random list and each patients' code will be kept in an opaque sealed envelope. Patients will be randomly allocated with 1:1 allocation ratio into two groups in a parallel manner:

* Group A: Patients will be managed using the modified pull-out suture technique.
* Group B: Patients will undergo repair using mini suture anchors.

  - Inclusion Criteria:
* Patients aged 18-55 years.
* Both sexes.
* Isolated volar plate injury.
* Closed injuries.
* Injury duration < 7 days.
* Willingness to participate and follow rehabilitation protocol.

  - Exclusion Criteria:
* Osteoprotic patients
* Associated neurovascular or tendon injuries.
* Open fractures or infections.
* Previous surgeries on the same finger.
* Inability to follow up.

ELIGIBILITY:
Inclusion Criteria::

* Patients aged 18-55 years.
* Both sexes.
* Isolated volar plate injury.
* Closed injuries.
* Willingness to participate and follow rehabilitation protocol.

Exclusion Criteria:

* Osteoprotic patients
* Associated neurovascular or tendon injuries.
* Open fractures or infections.
* Previous surgeries on the same finger.
* Inability to follow up.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
range of motion by geniometer | 6weeks